CLINICAL TRIAL: NCT03108300
Title: The Use of Propranolol Hydrochloride Combined With Anthracyclin Based Chemotherapy in the Treatment of Metastatic Soft Tissue Sarcoma
Brief Title: Use of Propranolol Hydrochloride in the Treatment of Metastatic STS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Nagy, Principal Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURE002
Record Dates: First submitted 2017-03-16; First posted 2017-04-11 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Malignant Soft Tissue Sarcoma
Keywords: efficacy; propranolol hydrochloride; sts
MeSH Terms: conditions — Ichthyosis, X-Linked | interventions — Propranolol; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- propranolol hydrochloride with Doxorubicin (Experimental): The patients suffering from metastatic soft tissue sarcoma will receive doxorubicin 60mg per square meter of body surface area every 21 days combined with propranolol hydrochloride 40mg twice daily
  Interventions: Drug: Propranolol Hydrochloride; Drug: Doxorubicin

INTERVENTIONS:
Drug: Propranolol Hydrochloride — propranolol hydrochloride is a beta-adrenergic receptor blocker
Drug: Doxorubicin — Doxorubicin is a chemotherapy which will be injected by a dose 60 mg per meter square of body surface area to be repeated every 21days
  Other Names: Adriamycin

SUMMARY:
Fifty patients with pathological proof of malignant soft tissue sarcoma will receive Anthracyclin based chemotherapy combined with propranolol 40 mg twice daily.

* The primary end point : To assess Progression Free Survival (PFS)
* The secondary end points : To assess Overall Survival (OS) and Toxicity Profile

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of malignant soft tissue sarcoma.
2. ECOG less than or equal to 2 .
3. Measurable disease according to the requirements of modified RECIST criteria.
4. Age ≥ 19 years .
5. Estimated life expectancy of at least 12 weeks .
6. Adequate bone marrow reserve (white blood cells [WBC] ≥ 3.5 × 109 /L, neutrophils ≥ 1.5 × 109 /L, platelets ≥ 100 × 109 /L, and hemoglobin ≥ 9.0 gm/dL).

Exclusion Criteria:

1. Inadequate liver function (bilirubin > 1.5 times upper normal limit [UNL] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3.0 UNL or up to 5.0 UNL in the presence of hepatic metastases).
2. Inadequate renal function (creatinine > 1.25 times UNL, creatinine clearance < 50mL/min).
3. Serious concomitant systemic disorder incompatible with the study.
4. Second primary malignancy (except in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior to enrollment without recurrence).
5. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | an average of 1 year
  Progression free survival (PFS) is defined as the time interval between the dates of first treatment administration and first observation of PD.

SECONDARY OUTCOMES:
Overall Survival | an average of 3 years
  Overall Survival (OS) is defined as the time from the date of the first treatment administration to the date of death due to any cause.

IPD SHARING:
Plan to Share IPD: No